CLINICAL TRIAL: NCT04329442
Title: Point of Care PrEP Delivery for Young Black/African American Men Who Have Sex With Men and Young Transgender Women at High Risk for HIV Infection
Brief Title: Accelerated PrEP Access for Black MSM and TW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 caused substantial barriers to recruitment.
Sponsor: University of Chicago (Other)
Collaborators: Planned Parenthood Great Plains (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB19-1154
Record Dates: First submitted 2020-03-26; First posted 2020-04-01 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: HIV/AIDS
Keywords: PrEP; HIV Prevention; Young Men Who Have Sex with Men; Young Transgender Women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: A single-arm longitudinal pre/post study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP Received (Experimental): Participants will be provided with a free 30-day supply of PrEP.
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet

INTERVENTIONS:
Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet — 30 day supply of 200mg tablets
  Other Names: Truvada

SUMMARY:
The investigators will pilot-test an accelerated PrEP initiation approach among young high-risk Black/African American (B/AA) men who have sex with men (MSM) and transgender women (YMSM/TW) at the point of care in community contexts.

DETAILED DESCRIPTION:
The study team will provide a free 30-day supply of HIV pre-exposure prophylaxis (PrEP) to young Black MSM and TW identified as PrEP-eligible and interested in taking PrEP to reduce their risk of HIV acquisition. This intervention is intended to assist youth at high risk for HIV acquisition in successfully initiating PrEP use.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-24;
2. assigned male at birth, identify as a man (cisgender), transgender woman, or gender non-conforming or genderqueer;
3. identifying as Black, African American, or multiracial with at least one parent identifying as Black or African American;
4. not currently taking PrEP or attending a visit to initiate PrEP;
5. self-report being HIV-negative;
6. reporting one of the following HIV risks in the last 6 months (Hosek, Rudy et al. 2015, Hosek, Rudy et al. 2017): a. condomless anal intercourse with an HIV-infected male partner or a male partner of unknown HIV status; b. anal intercourse with 3 or more male sex partners; c. exchange of money, gifts, shelter, or drugs for anal sex with a male partner; d. sex with a male partner and has had a sexually transmitted infection; e. sexual partner of an HIV-infected male with whom condoms were not consistently used; f. anal intercourse where the condom broke or slipped off

Exclusion Criteria:

* We are excluding those individuals who were assigned female at birth (female birth certificate) and/or cis-gender women (those assigned female at birth and identify as women) from the all phases of this study as this study is intended to explore the HIV prevention behaviors of B/AA young men who have sex with men and young transgender women (assigned male at birth) as these two groups represent the highest risk groups for HIV infection in the US, yet only a small percentage are aware or currently use PrEP for HIV prevention.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is open to cisgender men who have sex with men and transgender women.
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Intention to Continue PrEP | Post Intervention (1 month after receiving intervention)
  Intention to continue use of PrEP will be assessed via survey questions related to a respondent having made a follow-up appointment to continue taking PrEP, attended an appointment to continue taking PrEP, having filled a prescription for PrEP, and reporting an interest in continuing PrEP after current supply is complete.
Intention to Continue PrEP | Post Intervention (4 months after receiving intervention)
  Intention to continue use of PrEP will be assessed via survey questions related to a respondent having made a follow-up appointment to continue taking PrEP, attended an appointment to continue taking PrEP, having filled a prescription for PrEP, and reporting an interest in continuing PrEP after current supply is complete.
PrEP Adherence | Post Intervention (1 month after receiving intervention)
  PrEP adherence will be assessed via self-report of how many pills from the initial intervention remain and a self-assessment of success at remembering to take PrEP daily.
PrEP Adherence | Post Intervention (4 months after receiving intervention)
  PrEP adherence will be assessed via self-report of how many pills from the initial intervention remain and a self-assessment of success at remembering to take PrEP daily.

SECONDARY OUTCOMES:
PrEP Adherence Self-Efficacy | Post Intervention (1 month after receiving intervention)
  PrEP adherence self-efficacy will be assessed via a 9-question scale focused on respondents' belief that they could continue to take PrEP when experiencing barriers to adherence. Each item is scored on a 0-10 scale, where 0 means "cannot do at all" and 10 means "completely certainly can do." This scale has been adapted from the Adherence Self-Efficacy Scale (Johnson et al., 2007).
PrEP Adherence Self-Efficacy | Post Intervention (4 months after receiving intervention)
  PrEP adherence self-efficacy will be assessed via a 9-question scale focused on respondents' belief that they could continue to take PrEP when experiencing barriers to adherence. Each item is scored on a 0-10 scale, where 0 means "cannot do at all" and 10 means "completely certainly can do." This scale has been adapted from the Adherence Self-Efficacy Scale (Johnson et al., 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Darnell N Motley, PhD, Study Director — University of Chicago